CLINICAL TRIAL: NCT00247377
Title: A Prospective Randomized Trial of Laparoscopic Gastric Bypass vs Laparoscopic Adjustable Gastric Banding (LAP-BAND) for Treatment of Morbid Obesity
Brief Title: Laparoscopic Gastric Bypass vs LAP-BAND for Treatment of Morbid Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Nihn Tuan Nguyen, Chair and Professor, Department of Surgery, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-2002-2394
Record Dates: First submitted 2005-10-31; First posted 2005-11-01 (Estimated); Results first posted 2010-04-06 (Estimated); Last update posted 2023-04-24 (Actual); Status verified 2023-03

CONDITIONS: Morbid Obesity
Keywords: Morbid Obesity; Laparoscopic Gastric Bypass; Laparoscopic Gastric Banding
MeSH Terms: conditions — Obesity, Morbid | interventions — Gastric Bypass; Coronary Artery Bypass; Bariatric Surgery; Chromosome Banding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laparoscopic Gastric Bypass (Active Comparator): Subject undergoes Laparoscopic Gastric Bypass
  Interventions: Procedure: Gastric bypass surgery
- LAP-BAND (Active Comparator): Subject undergoes LAP-BAND procedure
  Interventions: Procedure: Lap-Band

INTERVENTIONS:
Procedure: Gastric bypass surgery — in order to meet health requirements for patient, gastric bypass surgery was undergone
  Other Names: gastric bypass; bypass surgery; weight loss surgery
  Arms: Laparoscopic Gastric Bypass
Procedure: Lap-Band — in order to meet health requirements for patient, gastric band surgery was undergone
  Other Names: weight loss surgery; band
  Arms: LAP-BAND

SUMMARY:
PURPOSE Obesity is a growing problem in the United States. Severe obesity, known as "morbid obesity", is defined as being 100 pounds in excess of ideal body weight. Nonsurgical treatments for morbid obesity include exercise, dietary restriction, behavior modification, and pharmacological intervention. However, it is estimated that most patients undergoing nonsurgical treatments for weight reduction will regain their weight within 2 to 4 years after treatment. According to the NIH consensus conference in 1991, surgery remains the only effective sustained weight loss treatment for morbid obesity. The Roux-en-Y gastric bypass (GBP) is currently considered the gold standard bariatric surgical operation. Mean weight loss following GBP is approximately 65% of the excess body weight during the first 12 to 18 months postoperatively. Long-term weight loss is in the range of 55-70% of excess body weight loss.

Recently, the laparoscopic approach to GBP was reported. Wittgrove and colleagues reported their results of 75 patients who underwent laparoscopic GBP and demonstrated significant short-term advantages with comparable weight loss and reversal of comorbidities compared to the open approach. However, GBP might it be done laparoscopic or open approach can potentially be associated with significant morbidity and mortality such as anastomotic leak, pulmonary embolism, bowel obstruction, and postoperative stricture.

The FDA recently approved the laparoscopic adjustable banding system (LAP-BAND) for use in the United States in June 2001. The LAP-BAND system is a device designed to induce weight loss in severely obese patients. It is surgically placed around the proximal stomach to create a small proximal stomach pouch and restricted opening, or stoma, through which passage of food will be slowed. An inflatable portion along the inner aspect of the band is connected to an access port, placed intramuscularly. This enabled stoma adjustments to be made without the need for further surgery. The advantages of the LAP-BAND system included no cutting or opening of the stomach wall, ability to adjust the stoma and a technically easier operation to perform than laparoscopic GBP. We wanted to evaluate if the LAP-BAND procedure is as effective as the laparoscopic GBP procedure for treatment of morbid obesity.

DETAILED DESCRIPTION:
RATIONALE:

1. Morbid obesity and its health consequences is increasing in the United States
2. Roux-en-Y GBP is an effective treatment for morbid obesity but can be associated with substantial morbidities
3. LAP-BAND system can be an effective treatment for morbidly obese patients with potentially reduced morbidity compared to laparoscopic GBP

HYPOTHESIS:

1. LAP-BAND can be performed safely and are associated with reduced postoperative pain, decrease in morbidity, decrease ICU and hospital stay, reduced costs, comparable improvement in quality-of-life, and acceptable long-term weight loss compared with laparoscopic GBP
2. LAP-BAND is associated with a decrease in fluid requirement in the perioperative period, improved postoperative pulmonary function, and lower intraabdominal pressure compared to laparoscopic GBP
3. LAP-BAND does not alter esophageal motility and is effective in improvement of gastroesophageal reflux disease (GERD) symptoms.

OBJECTIVES AND SPECIFIC AIMS:

1. To determine the short-term outcome, quality-of-life, costs, and long-term weight loss after laparoscopic GBP compared with LAP-BAND.
2. To compare physiologic changes such as perioperative fluid requirement, postoperative pulmonary function, and intraabdominal pressure after laparoscopic GBP and LAP-BAND.
3. To evaluate the effect of LAP-BAND on esophageal motility and its effectiveness in controlling gastroesophageal reflux symptoms (GERD) for morbidly obese patients with GERD.

Please note: All physician, hospital, laboratory costs, the barium study tests, and the performance of the operation will be billed to the subject or their insurer as customary since these procedures are standard of care regardless of participation in the study. The research procedures such as the pulmonary function tests, intra-abdominal pressure, body fat composition tests, resting energy expenditure, exercise testing, strength testing, nutritional assessments, and esophageal function tests are considered research-related and will be paid for by the investigator.

ELIGIBILITY:
Eligibility:

Inclusion Criteria:

1. Male or female patients with BMI of 40-60 kg/m2 or 35 kg/m2 with comorbidities
2. Good health status with acceptable operative risk (good cardiopulmonary function)
3. Willingness to follow protocol requirements: Signing informed consent, follow-up, and completing protocol diagnostic tests

Exclusion Criteria:

1. Prior upper abdominal surgery except cholecystectomy
2. Large abdominal ventral hernia
3. Patients with hiatal hernia
4. Inadequate prior medical management
5. Lack of patient's motivation and contribution to long-term success
6. Unacceptable operative risk
7. Minors and pregnant women are excluded as these patients do not qualify for the bariatric procedures. Minors are not psychologically fit to undergo such surgery and pregnant women are excluded because of safety for the fetus.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 197 (Actual)
Dates: Start 2002-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ninh T Nguyen, MD, Principal Investigator — University of California, Irvine Medical Center, Orange, CA
Locations (1):
- Univeristy of California, Irvine, Medical Center, Orange, California, United States

REFERENCES:
- [Result] Nguyen NT, Slone JA, Nguyen XM, Hartman JS, Hoyt DB. A prospective randomized trial of laparoscopic gastric bypass versus laparoscopic adjustable gastric banding for the treatment of morbid obesity: outcomes, quality of life, and costs. Ann Surg. 2009 Oct;250(4):631-41. doi: 10.1097/SLA.0b013e3181b92480. PMID 19730234
- See also: PubMed Abstract — http://www.ncbi.nlm.nih.gov/pubmed/19730234?itool=EntrezSystem2.PEntrez.Pubmed.Pubmed_ResultsPanel.Pubmed_RVDocSum&ordinalpos=2

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment between 2002 and 2007 in our bariatric surgery clinic
Pre-assignment Details: Patients were excluded because they did not want to undergo the randomized assignment or inability to obtain insurance coverage for the operation
Groups:
- Laparoscopic Gastric Bypass: Laparoscopic Gastric Bypass instead of LAP-Band
- Laparoscopic Adjustable Gastric Banding (LAP-BAND): Laparoscopic Adjustable Gastric Banding (LAP-BAND)instead of laparoscopic gastric bypass
Period: Overall Study
Arm/Group | Laparoscopic Gastric Bypass | Laparoscopic Adjustable Gastric Banding (LAP-BAND)
Started | 111 | 86
Completed | 111 | 86
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Laparoscopic Gastric Bypass | Laparoscopic Adjustable Gastric Banding (LAP-BAND) | Total
Number analyzed (Participants) | 111 | 86 | 197
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 111 | 86 | 197
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (11.0) | 45.8 (9.8) | 43.6 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 65 | 151
  Male | 25 | 21 | 46
Region of Enrollment [Number; unit: participants]
  United States | 111 | 86 | 197

OUTCOME MEASURES:

1. Secondary Outcome: Changes in Quality of Life- Physical Functioning Using SF-36 Questionnaire Pre-operation to 12 Months Post-operation
Description: change in quality of life survey response where 0 is non-functioning and 100 is fully functioning
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Laparoscopic Gastric Bypass | Laparoscopic Adjustable Gastric Banding (LAP-BAND)
Number analyzed (Participants) | 111 | 86
units on a scale | 86.8 (14.2) | 93.1 (8.8)

2. Primary Outcome: Excess Weight Loss From Pre-operation to 5 Years Post-operation
Description: weight loss as measured by change in percent of excess body weight
Time Frame: Baseline to 5 years
Population: Availability of subjects and protocol design
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Laparoscopic Gastric Bypass | Laparoscopic Adjustable Gastric Banding (LAP-BAND)
Number analyzed (Participants) | 111 | 86
percent change | 68.4 (19.5) | 45.4 (27.6)

3. Secondary Outcome: Cost of Procedure to the Medical Facility on Date of Procedure
Description: operative and post-operative direct costs including hospital service costs per patient. costs reflect the average cost per patient in each of the two groups (band vs. bypass) at a single time point: date of surgery.
Time Frame: date of surgery
Measure: Mean (Standard Deviation); unit: dollars per patient
Arm/Group | Laparoscopic Gastric Bypass | Laparoscopic Adjustable Gastric Banding (LAP-BAND)
Number analyzed (Participants) | 111 | 86
dollars per patient | 12310 (3099) | 10767 (1631)

4. Secondary Outcome: Changes in Quality of Life- Role- Physical Using SF-36 Questionnaire Pre-operation to 12 Months Post-operation
Description: change in quality of life survey response for physical aspects of life using the SF-36 questionnaire where 0 corresponds to no Role-Physical and 100 corresponds to full Role-Physical
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Laparoscopic Gastric Bypass | Laparoscopic Adjustable Gastric Banding (LAP-BAND)
Number analyzed (Participants) | 111 | 86
units on a scale | 88.2 (12.5) [0 to 100] | 100.0 (0) [0 to 100]

5. Secondary Outcome: Changes in Quality of Life- Bodily Pain Using SF-36 Questionnaire Pre-operation to 12 Months Post-operation
Description: change in quality of life survey response for bodily pain using the SF-36 questionnaire where 0 corresponds to no bodily pain and 100 corresponds to complete bodily pain
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Laparoscopic Gastric Bypass | Laparoscopic Adjustable Gastric Banding (LAP-BAND)
Number analyzed (Participants) | 111 | 86
units on a scale | 81.1 (28.8) | 84.5 (24.5)

6. Secondary Outcome: Changes in Quality of Life: General Health Using SF-36 Questionnaire Pre-operation to 12 Months Post-operation
Description: change in quality of life survey response for general health using the SF-36 questionnaire where 0 corresponds to no general health satisfaction and 100 corresponds to complete health satisfaction
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Laparoscopic Gastric Bypass | Laparoscopic Adjustable Gastric Banding (LAP-BAND)
Number analyzed (Participants) | 111 | 86
units on a scale | 82.7 (18.1) | 85.3 (12.7)

7. Secondary Outcome: Changes in Quality of Life- Vitality Using SF-36 Questionnaire Pre-operation to 12 Months Post-operation
Description: change in quality of life survey response for vitality as measured using the SF-36 questionnaire with worst score being 0 and best score being 100 on a 1-100 point scale.
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Laparoscopic Gastric Bypass | Laparoscopic Adjustable Gastric Banding (LAP-BAND)
Number analyzed (Participants) | 111 | 86
units on a scale | 73.2 (22.4) | 71.3 (14.3)

8. Secondary Outcome: Changes in Quality of Life- Social Functioning Using SF-36 Questionnaire Pre-operation to 12 Months Post-operation
Description: change in quality of life survey response for social functioning as measured using the SF-36 questionnaire where 0 corresponds to no social functioning and 100 corresponds to full social functioning
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Laparoscopic Gastric Bypass | Laparoscopic Adjustable Gastric Banding (LAP-BAND)
Number analyzed (Participants) | 111 | 86
units on a scale | 92.8 (12) | 81.3 (31.3)

9. Secondary Outcome: Changes in Quality of Life- Role- Emotional Using SF-36 Questionnaire Pre-operation to 12 Months Post-operation
Description: change in quality of life survey response for the emotional role using the SF-36 questionnaire where 0 corresponds to no emotional role and 100 corresponds to full emotional role
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Laparoscopic Gastric Bypass | Laparoscopic Adjustable Gastric Banding (LAP-BAND)
Number analyzed (Participants) | 111 | 86
units on a scale | 82.5 (47.6) | 100 (0)

10. Secondary Outcome: Changes in Quality of Life- Mental Health Using SF-36 Questionnaire From Pre-operation to 12 Months Post-operation
Description: change in quality of life survey response for mental health using the SF-36 questionnaire where 0 corresponds to no mental health well-being and 100 corresponds to complete mental health well-being
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Laparoscopic Gastric Bypass | Laparoscopic Adjustable Gastric Banding (LAP-BAND)
Number analyzed (Participants) | 111 | 86
units on a scale | 83.6 (14.1) | 86 (14.3)

ADVERSE EVENTS:
Time Frame: 2002-2007
Arm/Group | Laparoscopic Gastric Bypass | Laparoscopic Adjustable Gastric Banding (LAP-BAND)
Serious Adverse Events (participants affected / at risk) | 36/111 | 12/86
Other Adverse Events (participants affected / at risk) | 32/111 | 4/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Laparoscopic Gastric Bypass (N=111) | Laparoscopic Adjustable Gastric Banding (LAP-BAND) (N=86)
gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
gastrointestinal obstruction (Gastrointestinal disorders) | 4 (4) | 1 (1)
internal herniation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
anastomotic stricture (General disorders) | 17 (17) | 0 (0)
internal hernia (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
ventral hernia (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
death related to alcohol (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
marginal ulcer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
abdominal pain requiring laparoscopy (Gastrointestinal disorders) | 2 (2) | 0 (0)
bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
peripheral neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
renal insufficiency (Renal and urinary disorders) | 0 (0) | 1 (1)
anastomotic leak (Surgical and medical procedures) | 0 (0) | 0 (0)
port revision (Surgical and medical procedures) | 0 (0) | 3 (3)
band erosion/slippage erosion (Surgical and medical procedures) | 0 (0) | 5 (5)
failure of weight loss requiring revision of anastomosis (General disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Laparoscopic Gastric Bypass (N=111) | Laparoscopic Adjustable Gastric Banding (LAP-BAND) (N=86)
Dehydration require readmission (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 2 (3) | 1 (3)
Clinically significant atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 7 (7) | 0 (0)
Prolonged Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (2) | 1 (2)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Marginal ulcer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9) | 0 (0)
Gastrointestinal Bleeding (Gastrointestinal disorders) | 2 (2) | 0 (0)
Severe iron deficiency requiring iron infusion (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Alcohol Abuse (Social circumstances) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No